CLINICAL TRIAL: NCT05934578
Title: Lymphatic Function in Patients With Fontan Circulation: Effect of Physical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Copenhagen University Hospital, Denmark (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Aida Luiza R Turquetto, Principal investigator, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 61404222.6.0000.0068
Record Dates: First submitted 2022-11-17; First posted 2023-07-07 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Univentricular Heart; Congenital Heart Disease; Lymphatic Abnormalities; Functional Capacity; Exercise Training; Quality of Life
Keywords: Lymphatic dysfunction; Near-Infrared Fluorescence Imaging; Fontan circulation; Plethysmography; Functional capacity; Aerobic exercise; Cardiac rehabilitation; Capillary filtration; Exercise training
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital; Lymphatic Abnormalities | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A longitudinal clinical trial, controlled and no-randomized. Intervention: Exercise (aerobic and light muscle resistance exercise)
Who Masked: Outcomes Assessor
Masking Description: Two groups, one of them (10) will be submitted to an exercise program, and the other (10) will be maintained usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fontan Group - Exercise Training (Experimental): Online rehabilitation: 36 sessions of aerobic exercise training for two months
  Interventions: Other: Exercise training
- Fontan Control Group - No Exercise Training (No Intervention): Patients will not participate in the exercise program and will continue with their usual routine.

INTERVENTIONS:
Other: Exercise training — Aerobic and light muscle resistance exercise by online cardiovascular rehabilitation
  Arms: Fontan Group - Exercise Training

SUMMARY:
Background: The Fontan operation has been used to treat complex cardiac anomalies with a single-functioning ventricle. A study performed by Instituto do Coracão-Hospital das Clínicas-Universidade de Sao Paulo (InCor/HCFMUSP)-Brazil, Hospital das Clínicas of Ribeirão Preto-Brazil, department of the University of Aarhus, and Rigshospitalet, Denmark demonstrated an impairment peripheral lymphatic function in Fontan patients compared with healthy controls. However, the ability to increase the frequency of contractions is impaired when stressed by hyperthermia. Lymph vessels in Fontan patients were unable to respond usually. The participants were only able to increase the frequency of contraction twice during stress, compared to a five-fold increase among healthy controls. At the microcirculation level, Fontan patients filtered less fluid into the capillaries interstitial space than healthy controls at venous occlusion pressure. Studies carried out at InCor/HCFMUSP demonstrated that supervised aerobic exercise training improves the functional capacity and neurovascular control in Fontan patients compared to the non-training control group. However, the effect of aerobic exercise and light muscle resistance performed through online rehabilitation has not yet been demonstrated in peripheral lymphatic function and microcirculation. Aim: Evaluate the effects of an aerobic and light muscle resistance exercise program on peripheral lymphatic function, capillary filtration, functional capacity, and quality of life in adults with Fontan circulation. Methods: The function of the superficial lymphatic vessels in the lower leg will be investigated during rest in supine and standing positions, using near-infrared fluorescence imaging using Indocyanine Green (ICG; Verdye, Diagnostic Green GmbH, Germany). The variables analyzed are contraction frequency (contraction/minute), pumping Pressure (mmHg), and packet velocity. Venous congestion plethysmography will perform to analyze the capillary filtration and cardiopulmonary exercise test for functional capacity. The quality of life will be evaluated using the SF-36 Short-Form questionnaire. Expected results: the physical training improves peripheral lymphatic function, capillary filtration, functional capacity, and quality of life in patients with biventricular compared to the control group (no exercise training)

DETAILED DESCRIPTION:
The study population is patients submitted to Fontan operation to treat complex congenital heart disease (univentricular circulation), who are followed at InCor Heart Institute in Sao Paulo.

The investigators will perform all measures baseline and after 36 sessions of aerobic exercise and light resistance (exercise group) or after eight weeks in usual care (control group).

ELIGIBILITY:
Inclusion Criteria:

* Fontan circulation
* Age above 18 years
* Agreeing to participate in the study and signing the informed consent form.

Exclusion Criteria:

* Motor alterations make it impossible to perform the cardiopulmonary test
* Mental illness
* Syndromes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Assessing Peripheral Lymphatic Function Using Near-Infrared Fluorescence Imaging: Contraction Frequency Analysis over a 6-Minute Baseline | After 8 weeks of exercise training program or usual rotine
  Change in peripheral lymphatic function will be evaluated by Near-Infrared Fluorescence Imaging expressed by Contraction frequency (minute-1). A contraction was defined as a visual validation of a packet moving through a Regions of interests (ROI) placed on each measurable vessel and/or increase in the intensity signal displayed in the LabVIEW program. Contractions were counted over the obtained 6-min baseline.
Quantifying Peripheral Lymphatic Function through Near-Infrared Fluorescence Imaging: Assessment of Packet Velocity (cm/s) between ROIs. | After 8 weeks of exercise training program or usual rotine
  Change in peripheral lymphatic function will be evaluated by Near-Infrared Fluorescence Imaging expressed by Packet velocity (cm/s). Two ROIs were placed 5-10 cm apart on each vessel in the baseline sequence. Packages moving continuously through both ROIs were included in the calculations. The distance between the two ROIs was divided by the time difference between the packet passing each ROI.
Assessing Peripheral Lymphatic Function through Near-Infrared Fluorescence Imaging: Determination of Pumping Pressure (mmHg). | After 8 weeks of exercise training program or usual rotine
  Change in peripheral lymphatic function will be evaluated by Near-Infrared Fluorescence Imaging expressed by Pumping pressure (mmHg). Pumping pressure was determined by occluding lymphatic vessels using a Hokanson sphygmomanometer cuff (Marcom Medical Denmark). A tourniquet was placed distally to the sphygmomanometer cuff to prevent any lymphatic flow and allowing manual emptying of the lymphatic vessels under and above the cuff, which be inflated to 80 mm Hg (Hokanson E20 Rapid cuff inflator, Hokanson AG101 air source, SC10 cuff; Marcom Medical, Denmark) and the tourniquet was released allowing lymph flow up to the distal border of the cuff. Then, the cuff pressure was reduced with 5 mm Hg every 5th min until the fluorescent dye passed under the inflated cuff at which point the reached pressure level was noted as the pumping pressure.

SECONDARY OUTCOMES:
Assessment of Capillary Filtration Rate Using Venous Occlusion Plethysmography | After 8 weeks of exercise training program or usual rotine
  The capillary filtration rate (CFR) can be evaluated using venous occlusion plethysmography. CFR is measured using a strain gauge plethysmography setup (Hokanson EC6 and E20; Marcom Medical, Denmark) connected to a PC via an analog-to-digital converter (ADInstruments, UK). The measurements were analyzed using Labchart 7 software.
  The procedure involves placing a cuff around the right calf, conducting venous congestion applying pressures ranging from 20 to 70 mm Hg each 3 min. A strain gauge was placed on the widest circumference of the calf to record an increase in volume.
  The CFR was measured as the slope of the time-volume change (%) curve at a steady state at the end of each pressure phase. Measurements were taken at 10 mm Hg pressure intervals from 20 to 70 mm Hg.
Functional capacity assessment 1 | After 8 weeks of exercise training program or usual rotine
  Change in functional capacity will be performed by cardiopulmonary exercise test and will be expressed by Peak VO2 (mL/kg/min). After the training program, an increase in the peak VO2 value between 5 to 10% is expected in relation to the baseline value
"Functional Capacity Assessment through Cardiopulmonary Exercise Test: Predicted Peak VO2 (%) as an Indicator of Training Program Effectiveness | After 8 weeks of exercise training program or usual rotine
  Change in functional capacity will be performed by cardiopulmonary exercise test and will be expressed by Predicted Peak VO2 (%). After the training program, an increase in the predicted peak VO2 value between 5 to 10% is expected in relation to the baseline value.
Assessment of Quality of Life Using Short Form 36 Questionnaire: A Multi-Domain Analysis with Scores Ranging from 0 to 100 | After 8 weeks of exercise training program or usual rotine
  Changes in quality of life will be measure by Short Form 36 questionnaire by 8 domains: Physical functioning, Physical role functioning, body pain, general health, vitality, social functioning, emotional role functioning, mental health. The quality of life classification for each domain is typically measured on a scale of 0 to 100, where a score close to 100 indicates a higher or superior quality of life, while a score near 0 suggests a lower or poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Coracao, Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo, Brazil